CLINICAL TRIAL: NCT05546424
Title: EMRESERVA A Program to Enhace Cognitive Reserve in Patients With Multiple Scleorisis
Brief Title: EMRESERVA to Enhance Cognitive Reserve in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: EMRESERVA
Record Dates: First submitted 2022-05-12; First posted 2022-09-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Change

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: Non-specific cognitive exercises included general advice from MS neuropsychologist specialists on how to manage cognitive difficulties and general cognitives exercises to improve cognitive performance elaborated at our MS Unit, using exercises like sudokus, crosswords and labyrinths.
  This control group will require the completion of at least 30 minutes of cognitive exercises daily from Monday to Friday for 5 months. As a complement, patients will be instructed to read newspapers or magazines at least 15 minutes daily.
  Interventions: Behavioral: EMRESERVA
- Intervention EMRESERVA: Specific cognitive rehabilitation program "EM-Reserva" will be provided by two specialized MS
  Neuropsychologists in groups of 6 participants who will meet approximately an hour weekly, for 5 months."EM reserva" cognitive program includes the following activities:
  1. Cognitive leisure tasks
  2. Physical exercises (workout exercises)
  3. Activities that promote social relationships (social exercises)
  Interventions: Behavioral: EMRESERVA

INTERVENTIONS:
Behavioral: EMRESERVA — training program will be carried out in groups (up to 6 patients) who will meet one hour once a week for 5 months.

SUMMARY:
Multiple Sclerosis(MS) is an immunological degenerative disease that affects central nervous system causing cognitive impairment, which is one of the most disabling symptoms in MS. Cognitive reserve may influence manifestations of symptoms of cognitive impairment in MS patients and could justify interindividual differences. Cognitive reserve hypothesis raises that enriching life experiences creates a higher capacity and efficiency of neural networks and protects against cognitive decline in neurological diseases.

Scientific evidence demonstrates that older adults with a higher educational,occupational attainment or engagement in cognitively stimulating leisure activities have a reduced risk of dementia.Systematic reviews report little efficacy of pharmacological and behavioral treatments impairment in cognitive functions in MS patients . As such, best treatment of cognitive impairment in MS may be a proactive prevention of cognitive decline in first place Through the application of the EM-Reserva program our goal is to evaluate if it is possible to improve cognitive skills of patients with MS without cognitive impairment versus those who undergo non-specific cognitive exercises. In the short and medium term, EM-Reserva program could improve cognitive performance and delay the appearance or modulate the severity of cognitive impairment in the course of the disease

DETAILED DESCRIPTION:
The cognitive profile is homogeneous in MS. This neuropsychological profile is characterised by impairment of memory ,speed of information processing, attention and executive functions. Periodic cognitive explorations are necessary to assess evolution of patients with MS. This evaluation helps to establish a neuropsychological profile which could help to study cognitive and emotional symptoms of MS. Therefore, using reliable cognitive tests could enable to study neuropsychological disorders associated with MS.

Impact of cognitive impairment on daily routine of people with MS can be diverse and is one of major causes of disability in MS. Therefore is vital to stablished which is the role of cognitive and brain reserve and if they could explain inconsistency between structural damage and cognitive functions in MS.

Attention, information processing speed, working memory, and verbal fluency have a positive impact in cognitive reserve. Therefore, our goal is to assess whether EM-Reserva specific cognitive program have a positive impact in these cognitive functions and maybe could prevent onset of cognitive impairment.

According to Sumowski and Leavitt three activities have a strong association with enhancement of cognitive reserve.

1. Cognitive leisure tasks These activities are 1) reading books, 2) reading magazines or newspapers, 3) producing art (for example, painting, poetry or sculpture), 4) writing non-art productions (for example, a newspaper or a blog), 5) playing a musical instrument, 6) playing structured games (for example, cards, board games, crossword puzzles) and 7) engaging in hobbies (for example, gardening, model building and web design).
2. Aerobical physical exercises
3. Activities that promote social relationships.Gatz and Sumowskihighlighted that the establishment of complex cognitive activities in daily life may be relevant in order to achieve a positive impact in cognitive reserve and delay the onset of cognitive symptoms.

Therefore, is proposed to evaluate cognitive impact of the "EMReserva" specific cognitive training to maintain or improve cognitive functions in patients with MS compared to a standard cognitive training. A five-month (20 weeks) intervention program is proposed to evaluate efficacy of cognitive training programs in patients with MS. Cognitive performance improvement has been found after 5-15 weeks (28-32) of cognitive training. On the other hand, musical techniques had been used in cognitive rehabilitation for 24-36 weeks (33-36)

OBJECTIVES(enter elsewhere) METHODS(enter elsewhere) This is a pragmatic, unicentric, observer-blinded Randomized Controlled Trial (RCT) comparing cognitive rehabilitation programme EM-Reserva (intervention) with usual cognitive care alone(control).

This trial will be conducted in Multiple Sclerosis Unit of Virgen Macarena Universitary Hospital (UEMAC) in Seville, Spain.

Neuropsychologists will check participants' availability to attend groups. Groups of 6 participants who could potentially attend for treatment at the same time and venue were individually randomized to either "EM-Reserva'' intervention or usual cognitive care on a 1:1 ratio. Allocation will be stratified by results of Cognitive Reserve Questionnaire.

Normative data of the CRC were determined using quartiles. In this way, a score equal to or less than 6 points, which belongs to quartile 1 (≤ C1), would place the subject's degree of cognitive reserve in the lower range. Between 7 and 9 points (C1-C2) would correspond to a cognitive reserve located in the medium-low range, while between 10 and 14 (C2-C3) would be considered mediumhigh.

Those scores ≥ 15 points would be classified as a cognitive reserve located in the upper category (≥ C4) (23) The allocation algorithm was held on a secure server using an Internet Based randomization system to obtain treatment allocations for each participant and will be stratified taking in account CRC Quartiles in order to avoid a selection bias. Neuropsychologists and participants will be aware of the group allocation. Neurologists will be blinded to group allocation and will perform SDMT (primary endpoint of the study) Non-specific cognitive exercises included general advice from MS neuropsychologist specialists on how to manage cognitive difficulties and general cognitives exercises to improve cognitive performance elaborated at our MS Unit, using exercises like sudokus, crosswords and labyrinths.

This control group will require completion of at least 30 minutes of cognitive exercises daily from Monday to Friday for 5 months. As a complement, patients will be instructed to read newspapers or magazines at least 15 minutes daily.

Specific cognitive rehabilitation program "EM-Reserva" will be provided by two specialized MS Neuropsychologists in groups of 6 participants who will meet approximately an hour weekly, for 5 months. "EM reserva" cognitive program includes the following activities:

1. Cognitive leisure tasks 1) Reading books. 2) Reading magazines or newspapers daily. 3) Creative tasks type "Zentagle" drawing, 1 production per week. 4) Writing non-artistic productions: Journal writing or summaries of weekly activities will be recommended. 5) Playing a musical instrument: weekly group piano lessons will be held with a piano keyboard. 6) Playing structured games: Weekly groups will be held to play board games. 7) Participate in socio-cultural activities such as museum visits, exhibitions, etc., once a month.
2. Physical exercises (workout exercises): Group workout will be carried out through a virtual platform three times a week (one hour per session) assisted by a specialized MS Neurophysioterapist.
3. Activities that promote social relationships (social exercises): through group piano teaching lessons, board games for groups and other group activities.

The "EM Reserva" cognitive training program will be carried out in groups (up to 6 patients) who will meet one hour once a week for 5 months. In addition, patients will perform 30 minutes of individual cognitive exercises at home from Monday to Friday (musical exercises with piano/reading/writing...) Physical exercises will be done using a virtual platform, conducted by a non-blinded Neurophysioterapist specialized in MS. Attendance and compliance will be recorded in both intervention/control groups. If participants missed a group session, they could attend early for the following session to catch up on the content they had missed.

Compliance with prescribed homework will also be evaluated and recorded. Outcomes assessed at 6 and 12 months after randomization included the SDMT, Brief Repeatable Battery of Neuropsychological Test (BRB-N), Vocabulary WAIS-IV, TMT A/B, WMI WAIS-IV, Tower of London test, phonetic and semantic fluencies (COWAT), MSQOL-54, BDI and BAI and PDQ-5.

Questionnaires will be administered by specialized MS Neuropsychologists. EDSS, number of relapses, number of new/enlarged T2 lesions on cerebral MRI and concomitant medications will also be recorded. This information will be collected by specialized MS Neurologists blinded to intervention (visit 0 and visit 12 months).

Study Assessments A specific Cognitive Battery of recognized validity and reliability in this type of patients is used for this purpose. Patients will perform Brief Repeatable Neuropsychological Test Battery for MS (BRB-N), which evaluates verbal and visual memory, attention, information processing speed and prefrontal functions.Other test such as buschke Selective Reminder test (SRT), 10/36 Spatial recall Test (10/36 SRT),Symbol Digit Modalities Test (SDMT), Paced Auditory serial addition task (PASAT) and Verbal fluency test (FV) and Trail Making Test A-B (TMT A-B) will be also perform.

To asses executive functions other tests will be used, such as Working Memory Index test (WAIS-IV),Tower of London,Controlled Oral Word Association Test (COWAT),Wechsler Abbreviated Intelligence Scale, Cognitive Reserve Questionnaire (CRQ).

In order to evaluate the effect of the programme quality of life test all patients will perform Multiple Sclerosis International Quality of Life questionnaire (MusiQoL-54) ,PDQ (Perceived Deficit Questionnaire), Modified fatigue impact scale (MFIS-5) and The Beck Depression Inventory (BDI)

WORK PLAN

1. To select 58 patients who met inclusion/exclusion criteria (VISIT 0). They will be randomized in two groups (Intervention/Control) and stratified taking in account the punctuation in Cognitive Reserve Questionnaire and age, in a randomized 1:1 masked manner.
2. VISIT 1 (+/- 3m from VISIT 0), evaluate cognitive performance in both groups, using SDMT, (form2), Vocabulary WAIS-IV, TMT A/B, WMI WAIS-IV, TLT, Tower of London test, phonetic and semantic fluencies (COWAT).Administer MSQOL-54, BDI and BAI and PDQ-5 tests.
3. VISIT 2 (6 m +/- 1 month) evaluate cognitive performance in both groups, using SDMT(Form 3), BRB-N (Form B) , Vocabulary WAIS-IV, TMT A/B, WMI WAIS-IV, TLT, Tower of London test, phonetic and semantic fluencies (COWAT). Administer MSQOL-54, BDI and BAI and PDQ-5 tests.
4. VISIT 3(12 m +/- 1 month) evaluate cognitive performance in both groups with SDMT (Form 1), BRB-N (Form A) , Wechsler Intelligence Scale Vocabulary subtest (WAIS IV), TMT A-B, work memory index (WAIS), Tower of London test, phonetic and semantic fluencies, and MSQOL-54.

   * Differences in neuropsychological tests before and after cognitive rehabilitation will be evaluated by ANOVA two-factors with replication adn Wilks' Lambda test to test the hypothesis of equality.

Each test performance will be adjusted by age, education, and gender.

- Clinical/demographic data will be assessed in visit 0, visit 2 and visit 3, including sex, age, time of MS evolution, number of relapses, Kurtzke's Expanded Disability Status Scale (EDSS), number of cerebral magnetic resonance T2 lesions and gadolinium enhanced lesions and if they are receiving any Disease Modifying treatment.

EXPECTED OUTCOMES Intellectual enrichment is associated with greater protective efficiency of manifestations of cognitive dysfunctions.

After administration of EMReserve program, cognitive improvement with enrichment of cognitve reserve is expected. This fact may be reflected in neuropsychological assessment scores of patients who were included in the program whereas measures of patients who undergo non-specific program will not be increased.

Patients who complete the EMReserva program, due to increased cognitive reserve, will be less likely to develop cognitive impairment at one year from baseline.

If the EMReserva program proves to be effective in improving cognitive capacities involved in cognitive reserve, it would be considered necessary to maintain these cognitive habits throughout life. Therefore, the mental, physical and social exercises based on this program would be implemented as part of the global approach to their disease.

The present study aims to invest resources in prevention of cognitive impairment in patients affected by MS given its high prevalence and the impact on their daily life and quality of life as they are a young working population with high mental demands.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years (both inclusive).
* Relapsing-remitting Multiple Sclerosis (RRMS) according to the 2017 McDonald Revised Criteria with less than 15 years of evolution.
* Patients with EDSS <3
* No cognitive impairment on the Brief Neuropsychological Battery of Rao (BRB-N) (Form A) corrected for age and education performed on the last three months in the MS Unit of Hospital Virgen Macarena (UEMAC) according to Amato´s criteria
* Able to attend group sessions.
* Patients able to give written Informed Consent.

Exclusion Criteria:

* Diagnosis of Secondary Progressive or Primary Progressive MS according to McDonald revised criteria (2017)
* No evidence of relapse or corticosteroid treatment in the 3 months prior to study inclusion.
* Had vision or hearing problems, such that they were unable to complete the cognitive assessments.
* Had concurrent severe medical or psychiatric conditions, which prevented them from engaging in treatment and/or Beck Depression Inventory > 20.
* Involved in other psychological intervention trials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients under follow-up in the Multiple Sclerosis unit, diagnosed with RRMS (according to the revised McDonald 2017 criteria) and without cognitive impairment will be selected. The presence or absence of cognitive impairment will be determined according to Amato´s criteria, and defined as the absence of a failure on at least two BRB-N tests, with scores of at least 1.5 SD below the scores of healthy controls
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Symbol Digit modality test | at month 6
  Change in mean scores. Asociate display symbol to corresponding number. Number of correct responses in 90 seconds

SECONDARY OUTCOMES:
Change in Trail Making Test form A and B | at 6 and 12 months.
  change in mean scores
Change in BRB-N subtest | at 6 and 12 months
  Change in mean scores
Change in Wechsler Intelligence Scale Vocabulary subtest (WAIS IV) mean scores at 6 and Change in Wechsler Intelligence Scale Vocabulary subtest (WAIS IV) mean scores at 6 and Change in Wechsler Intelligence Scale Vocabulary subtest | at 6 and 12 months
  Change in mean scores
Change in Work memory index (WAIS) | at 6 and 12 months
  Change in mean scores
Change in Tower of London test | at 6 and 12 months
  Change in mean scores
Change in Phonetic and semantic fluencies | at 6 and 12 months
  Change in mean scores
Change in Multiple Sclerosis Quality of Life-54 (MSQOL-54) questionnaire | at 6 and 12 months
  Change in mean scores
Change in Beck depression/anxiety questionnaires | at 6 and 12 months
  Change in mean scores
Change in MFIS-5 | at 6 and 12 months
  Change in mean scores
Change in Perceived Deficit Questionnaire (PDQ-5) | at 6 and 12 months
  Change in mean scores

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Pública Andaluza para la gestión de la Investigación en Salud de Sevilla (FISEVI), Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amato MP, Zipoli V, Portaccio E. Multiple sclerosis-related cognitive changes: a review of cross-sectional and longitudinal studies. J Neurol Sci. 2006 Jun 15;245(1-2):41-6. doi: 10.1016/j.jns.2005.08.019. Epub 2006 Apr 27. PMID 16643953
- [Result] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Result] Benedict RH, Cox D, Thompson LL, Foley F, Weinstock-Guttman B, Munschauer F. Reliable screening for neuropsychological impairment in multiple sclerosis. Mult Scler. 2004 Dec;10(6):675-8. doi: 10.1191/1352458504ms1098oa. PMID 15584493
- [Result] Schwartz CE, Snook E, Quaranto B, Benedict RH, Vollmer T. Cognitive reserve and patient-reported outcomes in multiple sclerosis. Mult Scler. 2013 Jan;19(1):87-105. doi: 10.1177/1352458512444914. Epub 2012 Apr 30. PMID 22546847
- [Result] Scarmeas N, Levy G, Tang MX, Manly J, Stern Y. Influence of leisure activity on the incidence of Alzheimer's disease. Neurology. 2001 Dec 26;57(12):2236-42. doi: 10.1212/wnl.57.12.2236. PMID 11756603
- [Result] Wilson RS, Mendes De Leon CF, Barnes LL, Schneider JA, Bienias JL, Evans DA, Bennett DA. Participation in cognitively stimulating activities and risk of incident Alzheimer disease. JAMA. 2002 Feb 13;287(6):742-8. doi: 10.1001/jama.287.6.742. PMID 11851541
- [Result] Verghese J, Lipton RB, Katz MJ, Hall CB, Derby CA, Kuslansky G, Ambrose AF, Sliwinski M, Buschke H. Leisure activities and the risk of dementia in the elderly. N Engl J Med. 2003 Jun 19;348(25):2508-16. doi: 10.1056/NEJMoa022252. PMID 12815136
- [Result] He D, Zhang Y, Dong S, Wang D, Gao X, Zhou H. Pharmacological treatment for memory disorder in multiple sclerosis. Cochrane Database Syst Rev. 2013 Dec 17;2013(12):CD008876. doi: 10.1002/14651858.CD008876.pub3. PMID 24343792
- [Result] Rosti-Otajarvi EM, Hamalainen PI. Neuropsychological rehabilitation for multiple sclerosis. Cochrane Database Syst Rev. 2014 Feb 11;2014(2):CD009131. doi: 10.1002/14651858.CD009131.pub3. PMID 24515630
- [Result] Sumowski JF. Cognitive Reserve as a Useful Concept for Early Intervention Research in Multiple Sclerosis. Front Neurol. 2015 Aug 20;6:176. doi: 10.3389/fneur.2015.00176. eCollection 2015. No abstract available. PMID 26347706
- [Result] Heaton RK, Nelson LM, Thompson DS, Burks JS, Franklin GM. Neuropsychological findings in relapsing-remitting and chronic-progressive multiple sclerosis. J Consult Clin Psychol. 1985 Feb;53(1):103-10. doi: 10.1037//0022-006x.53.1.103. No abstract available. PMID 3980815
- [Result] Potagas C, Giogkaraki E, Koutsis G, Mandellos D, Tsirempolou E, Sfagos C, Vassilopoulos D. Cognitive impairment in different MS subtypes and clinically isolated syndromes. J Neurol Sci. 2008 Apr 15;267(1-2):100-6. doi: 10.1016/j.jns.2007.10.002. Epub 2007 Nov 13. PMID 17997417
- [Result] Arnett P, Forn C. [Neuropsychological evaluation in multiple sclerosis]. Rev Neurol. 2007 Feb 1-15;44(3):166-72. Spanish. PMID 17285522
- [Result] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Result] Achiron A, Barak Y. Cognitive impairment in probable multiple sclerosis. J Neurol Neurosurg Psychiatry. 2003 Apr;74(4):443-6. doi: 10.1136/jnnp.74.4.443. PMID 12640060
- [Result] Deloire MS, Bonnet MC, Salort E, Arimone Y, Boudineau M, Petry KG, Brochet B. How to detect cognitive dysfunction at early stages of multiple sclerosis? Mult Scler. 2006 Aug;12(4):445-52. doi: 10.1191/1352458506ms1289oa. PMID 16900758
- [Result] Feuillet L, Reuter F, Audoin B, Malikova I, Barrau K, Cherif AA, Pelletier J. Early cognitive impairment in patients with clinically isolated syndrome suggestive of multiple sclerosis. Mult Scler. 2007 Jan;13(1):124-7. doi: 10.1177/1352458506071196. PMID 17294621
- [Result] Boringa JB, Lazeron RH, Reuling IE, Ader HJ, Pfennings L, Lindeboom J, de Sonneville LM, Kalkers NF, Polman CH. The brief repeatable battery of neuropsychological tests: normative values allow application in multiple sclerosis clinical practice. Mult Scler. 2001 Aug;7(4):263-7. doi: 10.1177/135245850100700409. PMID 11548987
- [Result] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Result] Amato MP, Prestipino E, Bellinvia A, Niccolai C, Razzolini L, Pasto L, Fratangelo R, Tudisco L, Fonderico M, Mattiolo PL, Goretti B, Zimatore GB, Losignore NA, Portaccio E, Lolli F. Cognitive impairment in multiple sclerosis: An exploratory analysis of environmental and lifestyle risk factors. PLoS One. 2019 Oct 21;14(10):e0222929. doi: 10.1371/journal.pone.0222929. eCollection 2019. PMID 31634346
- [Result] Nunnari D, De Cola MC, Costa A, Rifici C, Bramanti P, Marino S. Exploring cognitive reserve in multiple sclerosis: New findings from a cross-sectional study. J Clin Exp Neuropsychol. 2016 Dec;38(10):1158-67. doi: 10.1080/13803395.2016.1200538. Epub 2016 Jul 13. PMID 27410680
- [Result] Sumowski JF, Leavitt VM. Cognitive reserve in multiple sclerosis. Mult Scler. 2013 Aug;19(9):1122-7. doi: 10.1177/1352458513498834. PMID 23897894
- [Result] Rami L, Valls-Pedret C, Bartres-Faz D, Caprile C, Sole-Padulles C, Castellvi M, Olives J, Bosch B, Molinuevo JL. [Cognitive reserve questionnaire. Scores obtained in a healthy elderly population and in one with Alzheimer's disease]. Rev Neurol. 2011 Feb 16;52(4):195-201. Spanish. PMID 21312165
- [Result] Brickman AM, Siedlecki KL, Muraskin J, Manly JJ, Luchsinger JA, Yeung LK, Brown TR, DeCarli C, Stern Y. White matter hyperintensities and cognition: testing the reserve hypothesis. Neurobiol Aging. 2011 Sep;32(9):1588-98. doi: 10.1016/j.neurobiolaging.2009.10.013. Epub 2009 Nov 18. PMID 19926168
- [Result] Gatz M, Prescott CA, Pedersen NL. Lifestyle risk and delaying factors. Alzheimer Dis Assoc Disord. 2006 Jul-Sep;20(3 Suppl 2):S84-8. doi: 10.1097/00002093-200607001-00013. PMID 16917202
- [Result] Schwartz CE, Ayandeh A, Ramanathan M, Benedict R, Dwyer MG, Weinstock-Guttman B, Zivadinov R. Reserve-building activities in multiple sclerosis patients and healthy controls: a descriptive study. BMC Neurol. 2015 Aug 12;15:135. doi: 10.1186/s12883-015-0395-0. PMID 26264858
- [Result] Chiaravalloti ND, Moore NB, DeLuca J. The efficacy of the modified Story Memory Technique in progressive MS. Mult Scler. 2020 Mar;26(3):354-362. doi: 10.1177/1352458519826463. Epub 2019 Feb 11. PMID 30741103
- [Result] Mani A, Chohedri E, Ravanfar P, Mowla A, Nikseresht A. Efficacy of group cognitive rehabilitation therapy in multiple sclerosis. Acta Neurol Scand. 2018 Jun;137(6):589-597. doi: 10.1111/ane.12904. Epub 2018 Feb 7. PMID 29411360
- [Result] Bonavita S, Sacco R, Della Corte M, Esposito S, Sparaco M, d'Ambrosio A, Docimo R, Bisecco A, Lavorgna L, Corbo D, Cirillo S, Gallo A, Esposito F, Tedeschi G. Computer-aided cognitive rehabilitation improves cognitive performances and induces brain functional connectivity changes in relapsing remitting multiple sclerosis patients: an exploratory study. J Neurol. 2015 Jan;262(1):91-100. doi: 10.1007/s00415-014-7528-z. Epub 2014 Oct 12. PMID 25308631
- [Result] Vazquez-Marrufo M, Galvao-Carmona A, Gonzalez-Rosa JJ, Hidalgo-Munoz AR, Borges M, Ruiz-Pena JL, Izquierdo G. Neural correlates of alerting and orienting impairment in multiple sclerosis patients. PLoS One. 2014 May 12;9(5):e97226. doi: 10.1371/journal.pone.0097226. eCollection 2014. PMID 24820333
- [Result] Wan CY, Schlaug G. Music making as a tool for promoting brain plasticity across the life span. Neuroscientist. 2010 Oct;16(5):566-77. doi: 10.1177/1073858410377805. PMID 20889966
- [Result] Schellenberg EG. Music lessons enhance IQ. Psychol Sci. 2004 Aug;15(8):511-4. doi: 10.1111/j.0956-7976.2004.00711.x. PMID 15270994
- [Result] Bangert M, Altenmuller EO. Mapping perception to action in piano practice: a longitudinal DC-EEG study. BMC Neurosci. 2003 Oct 15;4:26. doi: 10.1186/1471-2202-4-26. PMID 14575529
- [Result] Herholz SC, Zatorre RJ. Musical training as a framework for brain plasticity: behavior, function, and structure. Neuron. 2012 Nov 8;76(3):486-502. doi: 10.1016/j.neuron.2012.10.011. PMID 23141061
- [Result] Moreno S, Marques C, Santos A, Santos M, Castro SL, Besson M. Musical training influences linguistic abilities in 8-year-old children: more evidence for brain plasticity. Cereb Cortex. 2009 Mar;19(3):712-23. doi: 10.1093/cercor/bhn120. Epub 2008 Oct 1. PMID 18832336
- [Result] Olivera-Souza RD, Moll J, Passman LJ, Cunha FC, Paes F, Adriano MV, Ignacio FA, Marrocos RP. Trail making and cognitive set-shifting. Arq Neuropsiquiatr. 2000 Sep;58(3B):826-9. doi: 10.1590/s0004-282x2000000500006. PMID 11018818
- [Result] Crowe SF. The differential contribution of mental tracking, cognitive flexibility, visual search, and motor speed to performance on parts A and B of the Trail Making Test. J Clin Psychol. 1998 Aug;54(5):585-91. doi: 10.1002/(sici)1097-4679(199808)54:53.0.co;2-k. PMID 9696108
- [Result] Shallice T. Specific impairments of planning. Philos Trans R Soc Lond B Biol Sci. 1982 Jun 25;298(1089):199-209. doi: 10.1098/rstb.1982.0082. PMID 6125971
- [Result] Staff RT, Murray AD, Deary IJ, Whalley LJ. What provides cerebral reserve? Brain. 2004 May;127(Pt 5):1191-9. doi: 10.1093/brain/awh144. Epub 2004 Mar 26. PMID 15047587
- [Result] Stanovich KE, Cunningham AE. Studying the consequences of literacy within a literate society: the cognitive correlates of print exposure. Mem Cognit. 1992 Jan;20(1):51-68. doi: 10.3758/bf03208254. PMID 1549065
- [Result] Sumowski JF, Chiaravalloti N, Wylie G, Deluca J. Cognitive reserve moderates the negative effect of brain atrophy on cognitive efficiency in multiple sclerosis. J Int Neuropsychol Soc. 2009 Jul;15(4):606-12. doi: 10.1017/S1355617709090912. PMID 19573279
- [Result] Aymerich M, Guillamon I, Perkal H, Nos C, Porcel J, Berra S, Rajmil L, Montalban X. [Spanish adaptation of the disease-specific questionnaire MSQOL-54 in multiple sclerosis patients]. Neurologia. 2006 May;21(4):181-7. Spanish. PMID 16832772
- [Result] Strober LB, Binder A, Nikelshpur OM, Chiaravalloti N, DeLuca J. The Perceived Deficits Questionnaire: Perception, Deficit, or Distress? Int J MS Care. 2016 Jul-Aug;18(4):183-90. doi: 10.7224/1537-2073.2015-028. PMID 27551243
- [Result] D'Souza E. Modified Fatigue Impact Scale - 5-item version (MFIS-5). Occup Med (Lond). 2016 Apr;66(3):256-7. doi: 10.1093/occmed/kqv106. No abstract available. PMID 27016749
- [Result] Goldman Consensus Group. The Goldman Consensus statement on depression in multiple sclerosis. Mult Scler. 2005 Jun;11(3):328-37. doi: 10.1191/1352458505ms1162oa. PMID 15957516